CLINICAL TRIAL: NCT01985438
Title: Prophylactic Nutritional Support During Treatment for Head and Neck Cancer: A Single-Center, Open-label, Prospective, Randomized, Controlled Trial Comparing Feeding With Percutaneous Endoscopic Gastrostomy Tubes and Nasogastric Tubes
Brief Title: A Trial Comparing Two Modalities of Prophylactic Nutritional Support During Treatment for Head and Neck Cancer
Acronym: PRONUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SKMCHRC-IRB-13-15
Record Dates: First submitted 2013-11-01; First posted 2013-11-15 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Head and Neck Neoplasms
Keywords: Head and Neck Neoplasms; Nutritional Support; Randomized Controlled Trial; Percutaneous Endoscopic Gastrostomy tube; Nasogastric tube; Radiation Effects; Pakistan
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- percutaneous endoscopic gastrostomy tube (Active Comparator): Percutaneous endoscopic gastrostomy tube placement - A 20 Fr PEG tube (Cook Medical, or Boston Scientific) will be placed endoscopically using Ponsky's pull technique, under conscious sedation, as a day-case procedure. A single dose of a prophylactic intravenous antibiotic (1.2g co-amoxiclav, 30 minutes prior to the procedure, unless evidence of penicillin allergy) will be given to all patients undergoing PEG tube insertion. Patients will be monitored for one hour prior to discharge following PEG tube insertion
  Interventions: Procedure: percutaneous endoscopic gastrostomy tube placement
- nasogastric tube (Active Comparator): Nasogastric tube placement - All nasogastric tubes will be inserted in a standard manner by a Gastroenterology Fellow or an Internal Medicine resident. Ordinarily, a 14 Fr, fine-bore NG feeding tube will be inserted at the bedside or, if unsuccessful, inserted under radiological guidance. A post-procedure abdominal x-ray will be performed to confirm correct placement of all NG tubes.
  Interventions: Procedure: nasogastric tube placement

INTERVENTIONS:
Procedure: percutaneous endoscopic gastrostomy tube placement — A 20 Fr PEG tube (Cook Medical, or Boston Scientific) will be placed endoscopically using Ponsky's pull technique, under conscious sedation, as a day-case procedure. A single dose of a prophylactic intravenous antibiotic (1.2g co-amoxiclav, 30 minutes prior to the procedure, unless evidence of penicillin allergy) will be given to all patients undergoing PEG tube insertion. Patients will be monitored for one hour prior to discharge following PEG tube insertion.
  Arms: percutaneous endoscopic gastrostomy tube
Procedure: nasogastric tube placement — All nasogastric tubes will be inserted in a standard manner by a Gastroenterology Fellow or an Internal Medicine resident. Ordinarily, a 14 Fr, fine-bore NG feeding tube will be inserted at the bedside or, if unsuccessful, inserted under radiological guidance. A post-procedure abdominal x-ray will be performed to confirm correct placement of all NG tubes.
  Arms: nasogastric tube

SUMMARY:
Purpose:

To compare the effect of prophylactic enteral feeding tube placement (either percutaneous endoscopic gastrostomy (PEG) tube or nasogastric (NG) tube) in patients undergoing treatment for head and neck cancer (HNC) on nutritional status, quality of life, mental and emotional health, rates of clinical complications, and cost of care.

Study Design:

Prospective randomized controlled trial with 2 arms and equal allocation ratio

Study Objectives:

1. The primary objective is to assess, among HNC patients randomized to receive either prophylactic PEG tube or NG tube for enteral support and who are undergoing chemo-radiation at SKMCH&RC, the change from baseline in nutritional status at the end of 24 weeks after treatment initiation.
2. The secondary objectives are to assess, among HNC patients randomized to receive either prophylactic PEG tube or NG tube for enteral support and who are undergoing chemo-radiation at SKMCH&RC, the change from baseline in nutritional status at the end of 12 weeks; the rates of complications; quality of life including symptoms of depression and anxiety; and cost of care (all related to enteral feeding tube placement only) at baseline and at the end of 12 weeks and 24 weeks after treatment initiation.

Patients and methods:

Eligible patients will be enrolled consecutively from the gastroenterology outpatient clinics at Shaukat Khanum Memorial Cancer Hospital and Research Center (SKMCH&RC), Lahore and randomly assigned to receive either PEG tube or NG tube placement prior to commencement of treatment. Patients will receive counseling from a trained nutritionist regarding adequate nutrition during treatment and enteral feeding tube care. Detailed information regarding demographics, cancer location, type and staging, clinical status, nutritional status, quality of life, mental and emotional health, and cost of care will be obtained at baseline (time at which cancer treatment is initiated) and on 21st day (3 weeks), 42nd day (6 weeks), 84th day (12 weeks) and 168th day (24 weeks) after initiating chemoradiation. The primary endpoint will be to compare the nutritional status between the two treatment groups on an intent-to-treat basis on 168th day (24 weeks) after initiating chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

* All treatment-naïve patients presenting to the Head and Neck outpatient Clinic at Shaukat Khanum Memorial Cancer Hospital and Research Centre, Lahore AND accepted into the system for treatment of a primary malignant neoplasm of head and neck (neoplasms of lip; oral cavity; pharynx; and larynx [see appendix for detailed definition and corresponding International Classification of Diseases 9th Revision Clinical Modification (ICD-9-CM) codes] AND referred to the Gastroenterology (GI) service for percutaneous endoscopic gastrostomy tube placement or nasogastric tube placement
* 18 years or older

Exclusion Criteria:

* Patients who have already received treatment for the neoplasm of head and neck at a center other than SKMCH&RC.
* Patients with recurrence following earlier treatment for cancer of the head and neck region.
* Patients presenting with neoplasms of nasal cavities, middle ear and accessory sinuses; skin of head, neck and face; neoplasms of eye; and neoplasms of brain.
* Patients with contraindications to PEG tube or NG tube placement.
* Patients with moderate to severe mental or physical disabilities because such disabilities will make it impossible to assess functional status deterioration related to the disease or its treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Nutritional Status | change from baseline nutritional status at 24 weeks after starting treatment
  Nutritional status will be assessed using three methods: (1) Patient-Generated Subjective Global Assessment (PG-SGA) tool, (2) anthropometric data, and (3) biochemical data. Biochemical assessment will be done by measuring serum albumin and electrolytes and kidney function tests. Primary outcome will be analyzed at aggregate level and after stratifying by age, sex, location of tumor, disease severity, and grade of dysphagia.

SECONDARY OUTCOMES:
Quality of Life + Mental/Emotional health | change from baseline quality of life & mental/emotional health scores at 12 and 24 weeks
  The quality of life will be assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) version 3.0. and Functional Assessment of Cancer Therapy Head and Neck (FACT H&N) version 4. Patients will also be assessed for their mental and emotional health. For this purpose, Hospital Anxiety and Depression Scale (HADS) will be used. All of these questionnaires are available in Urdu.
Cost of care | up to 24 weeks
  Data on cost of care associated with nutritional support will be assessed from the hospital's and patient's perspective.
Clinical Complications | up to 24 weeks
  Rate of minor and major clinical complications related to placement of PEG or NG tube will be assessed
Nutritional status | change in nutritional status from baseline at 12 weeks after starting treatment
  Nutritional status will be assessed using three methods: (1) Patient-Generated Subjective Global Assessment (PG-SGA) tool, (2) anthropometric data, and (3) biochemical data. Biochemical assessment will be done by measuring serum albumin and electrolytes and kidney function tests. All secondary outcomes will be analyzed at aggregate level and after stratifying by age, sex, location of tumor, disease severity, and grade of dysphagia.

CONTACTS AND LOCATIONS:
Overall Officials: M. Aasim Yusuf, MBBS, FRCP, Principal Investigator — Shaukat Khanum Memorial Cancer Hospital and Research Center; Waleed Zafar, MBBS, ScD, Principal Investigator — Shaukat Khanum Memorial Cancer Hospital and Research Center
Locations (1):
- Shaukat Khanum Memorial Cancer Hospital and Research Center, Lahore, Punjab Province, Pakistan